CLINICAL TRIAL: NCT00191308
Title: Molecular Profiling and Safety Study of Operable Lung Cancer Patients Treated With Alimta Combined With Cisplatin as Neoadjuvant Chemotherapy
Brief Title: Molecular Profiling in Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9356; H3E-PL-S051 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-04-20 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Non-Small Cell Lung Cancer; Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Pemetrexed; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Cisplatin (Experimental): Pemetrexed: 500 milligrams per square meter (mg/m^2) intravenous (IV) every 21 days (q 21 days) for 3 cycles unless disease progression occurs
  Cisplatin: 75 mg/m^2 IV q 21 days for 3 cycles unless disease progression occurs
  Interventions: Drug: pemetrexed; Drug: cisplatin; Procedure: Radical Non-Small Cell Lung Cancer (NSCLC) surgery

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m^2 IV q 21 days for 3 cycles unless disease progression occurs
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m^2 IV q 21 days for 3 cycles unless disease progression occurs
Procedure: Radical Non-Small Cell Lung Cancer (NSCLC) surgery — All participants proceeded to surgery within 4-8 weeks from the last dose of pemetrexed.

SUMMARY:
The main purpose of this study of pemetrexed combined with cisplatin used as neoadjuvant chemotherapy (2 or 3 cycles) in participants with operable non-small cell lung cancer (NSCLC) is to look at various genes present in participants' blood and tumor tissue to see if there is any link between the levels or changes in the genes and how participants with lung cancer respond to pemetrexed and cisplatin treatment.

ELIGIBILITY:
Inclusion Criteria:

* pathologic documentation of non-small cell lung cancer (NSCLC)
* tumor must be accessible by bronchoscopy for tumor tissue sample collection
* patients must have lung cancer with clinical stage IB, II, IIIA
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* patients must not have received prior systemic chemotherapy or radiation therapy for NSCLC (prior resection of lung is allowed provided at least 5 years have elapsed between prior surgery and enrolment)

Exclusion Criteria:

* bronchoalveolar carcinoma or stage IIIA tumor involving the superior sulcus (Pancoast tumors)
* pregnant or breast feeding patients
* patients who have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* patients with history or presence of other malignancy except in situ carcinoma of the skin or prior malignancy treated more than 5 years before without recurrence (excluding melanoma, breast cancer and hypernephroma)
* unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/ GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bystra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 500 milligram per square meter (mg/m^2) intravenous (IV) every 21 days (q 21 days) for 3 cycles unless disease progression occurs.
  Cisplatin: 75 mg/m^2 IV q 21 days for 3 cycles unless disease progression occurs.
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 30
Completed | 29
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 55.94 (8.214)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 30
Region of Enrollment [Number; unit: participants]
  Poland | 30
Basis for Diagnosis [Number; unit: participants]
  Histopathological | 30
  Cytological | 0
Initial Pathological Diagnosis [Number; unit: participants] — Pemetrexed was approved in April 2008 for first- and second-line treatment of locally advanced or metastatic non-small cell lung cancer (NSCLC), other than predominantly squamous. Of the 30 participants enrolled at that time, 20 had squamous cell histology. The protocol was not amended since enrollment stopped early (October 2008) due to lack of eligible participants.
  participants
    Adenocarcinoma of Lung | 2
    Mixed Cell Carcinoma of Lung | 0
    Squamous Cell Carcinoma of Lung | 20
    Large Cell Carcinoma of Lung | 0
    Bronchoalveolar Carcinoma | 0
    Other | 8
Stage of Disease at Study Entry [Number; unit: participants] — Tumor stages ranged from 0 (not spread) to IV (spread throughout the body). Stage IB=tumor was larger or grew deeper than IA, but was not in the lymph nodes; Stage IIA=cancer spread to some lymph nodes near the original tumor; Stage IIB=cancer was not in the lymph nodes but in the chest wall region, or was a larger tumor in the lymph nodes.
  participants
    Stage IB | 18
    Stage IIA | 2
    Stage IIB | 10

OUTCOME MEASURES:

1. Primary Outcome: High/Low Expression of Selected Molecular Markers in Tumor Tissues and Hypermethylated Genes in Peripheral Blood
Description: Molecular markers assessed by immunohistochemistry: thymidylate synthase, glycinamide ribonucleotide formyl transferase (GARFT), epidermal growth factor receptor (EGFR); and by polymerase chain reaction: dihydrofolate reductase (DHFR), dihydropyrimidine dehydrogenase (DPD), folylpolyglutamate synthetase (FPGS), reduced folate carrier, alpha folate receptor, Excision Repair Cross-Complementation Group 1 (ERCC1), folylpolyglutamate hydrolase (FPGH). Hypermethylated genes assessed by methylation-specific polymerase chain reaction. Due to small sample size, tumor-tissue analyses were not done.
Time Frame: Baseline, Cycle 2, and surgery (4-8 weeks after last dose of pemetrexed)
Population: Due to lack of eligible participants, enrollment was stopped early when 30 participants were enrolled. Tumor samples were collected in only 19 of these 30 participants. Results obtained from analyses of a small number of available samples were considered to be of little scientific and medical relevance, and tumor-tissue analyses were not conducted.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants With Objective Tumor Response (Response Rate)
Description: Tumor response to treatment using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=20% increase in sum of longest diameter of target lesions; Stable Disease (SD)=small changes that do not meet above criteria. Response rate was estimated as the total number of CR or PR, divided by the total number of participants treated.
Time Frame: Treatment start to disease progression or surgery (4-8 weeks after last dose of pemetrexed)
Population: Tumor response rate and 95% confidence interval (CI) of best CR or PR were evaluated on all qualified enrolled participants treated with at least 1 dose of study medication. Criteria=histological or cytological diagnosis of non-small cell lung cancer (NSCLC) IB-IIIA; presence of measurable disease; no previous NSCLC chemotherapy and radiotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 29
percentage of participants | 34.5 [17.9 to 54.3]

3. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time from complete response (CR) or partial response (PR) to disease progression. Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=20% increase in sum of longest diameter of target lesions.
Time Frame: Time of response to disease progression (up to 44.4 months)
Population: Duration of response was analyzed on responders treated with at least 1 dose of study medication. Criteria=histological or cytological diagnosis of non-small cell lung cancer (NSCLC) IB-IIIA; presence of measurable disease; no previous NSCLC chemotherapy and radiotherapy; responder.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 10
months | 42.5 [8.31 to NA] — The upper limit of the 95% confidence interval (CI) was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS was the time from date of first dose to first observation of progressive disease (PD) or death due to any cause. PD=20% increase in sum of longest diameter of target lesions. If a participant was not known to have died or have PD, DFS was censored at the date of the last objective progression-free disease assessment.
Time Frame: Treatment start to disease progression or death from any cause (up to 45.5 months)
Population: DFS was evaluated on all qualified enrolled patients who received at least 1 dose of study medication. Criteria=histological or cytological diagnosis of non-small cell lung cancer (NSCLC) IB-IIIA; presence of measurable disease; no previous NSCLC chemotherapy and radiotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 29
months | 43.7 [25.36 to NA] — The upper limit of the 95% confidence interval (CI) was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from treatment start to death from any cause. For participants who were alive, OS was censored at the last contact date.
Time Frame: Treatment start to death from any cause (up to 47.6 months)
Population: OS was evaluated on all qualified enrolled patients who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 29
months | NA [31.15 to NA] — The median and upper limit of the 95% confidence interval (CI) were not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=30)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=30)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Weight increased (Investigations) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Trial enrollment was terminated early due to lack of eligible participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days